CLINICAL TRIAL: NCT02619110
Title: The Purpose of This Study Was to Discuss on the Effects of Backward Walking Treadmill Training on Balance Ability, Speed of Walking and Cardiopulmonary Fitness for Patient With Chronic Stroke
Brief Title: The Effect of Backward Walking Treadmill Training on Balance in Patient With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KMUH-IRB-20130288
Record Dates: First submitted 2015-11-17; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-02

CONDITIONS: Stroke
Keywords: Chronic Stroke; cardiopulmonary; Berg Balance Scale (BBS)
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- backward walking treadmill training (Other): The intervention group not only received four weeks of conventional physical therapy but also accepted additional four weeks of backward walking treadmill training at the same time
  Interventions: Other: backward walking treadmill training; Other: conventional physical therapy
- conventional physical therapy (Other): The conventional physical therapy training focused on strengthening, postural control, functional mobility and forward gait training program but excluded backward walking training
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: backward walking treadmill training — subjects accepted 30 minutes backward walking treadmill training. a week for four weeks.
  Arms: backward walking treadmill training
Other: conventional physical therapy — subjects accepted 30 minutes traditional physical therapy three times a week for four weeks

SUMMARY:
The purpose of this research was to discuss the effect of backward walking treadmill training on balance ability, speed of walking and cardiopulmonary fitness in patients with chronic stroke.

DETAILED DESCRIPTION:
Walking training is a good method and strategy to improve postural stability, balance, gait symmetry, and increase walking ability. Generally, there are many walking training theories and methods for patients with chronic stroke and treadmill walking training is applied in recent years. Previous studies showed that patients with stroke improve the walking abilities and speed after the walking treadmill training. However, most studies have demonstrated that forward walking treadmill training improved balance and walking ability in patients with stroke, but fewer studies have investigated the effects on backward walking treadmill training. However, no studies to date have investigated the effects of backward walking treadmill training for patients with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* This experiment recruited subjects with chronic stroke more than six months, whose level of Brunnstrom stage was beyond IV and who were able to walk more than eleven meters with or without assistive devices

Exclusion Criteria:

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The change of Berg Balance Scale (BBS) | Baseline, week 4.

SECONDARY OUTCOMES:
The change of pulmonary function test (PFT): forced vital capacity (FVC) and Forced expiratory volume in one second (FEV1) | Baseline, week 4.

OTHER OUTCOMES:
Timed 10-Meter Walk Test (10 MWT) | 10 minutes
6-minute walk test (6 MWT) | 6-minute
Up and Go test (TUG) | Baseline, week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Y Guo, Ph.D, Study Chair — Department of Sports Medicine, College of Medicine, Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

REFERENCES:
- [Result] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS medicine 3(11):e442, 2006. Mendis S. Stroke disability and rehabilitation of stroke: World Health Organization perspective. International journal of stroke : official journal of the International Stroke Society 8(1):3-4, 2013 Chen CY, Huang YB, Tzu-Chi Lee C. Epidemiology and disease burden of ischemic stroke in Taiwan. The International journal of neuroscience 123(10):724-731, 2013 Bonita R, Beaglehole R. Recovery of motor function after stroke. Stroke; a journal of cerebral circulation 19(12):1497-1500, 1988 Niam S, Cheung W, Sullivan PE, Kent S, Gu X. Balance and physical impairments after stroke. Archives of physical medicine and rehabilitation 80(10):1227-1233, 1999
- [Derived] Chang KW, Lin CM, Yen CW, Yang CC, Tanaka T, Guo LY. The Effect of Walking Backward on a Treadmill on Balance, Speed of Walking and Cardiopulmonary Fitness for Patients with Chronic Stroke: A Pilot Study. Int J Environ Res Public Health. 2021 Mar 1;18(5):2376. doi: 10.3390/ijerph18052376. PMID 33804374